CLINICAL TRIAL: NCT05671172
Title: Effect of Adding Two Different Doses of Hyaluronidase to Bupivacaine in Ultrasound-Guided Transversus Abdominis Plane (TAP) Block for Post-cesarean Section Analgesia; A Randomized Controlled Double Blinded Study.
Brief Title: Effect of Adding Hyaluronidase to Bupivacaine in Transversus Abdominis Plane Block for Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, Doctor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC 4-8-2022
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Hyaluronoglucosaminidase; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group H1 (Experimental): patients will received TAB block with 19 ml bupivacaine 0.25 % plus 1 ml 0.9% normal saline containing 750 IU hyaluronidase as an adjuvant in each side after closing skin.
  Interventions: Drug: Hyaluronidase
- Group H2 (Experimental): patients will received TAB block with 19 ml bupivacaine 0.25 % plus 1 ml 0.9% normal saline containing 1500 IU hyaluronidase as an adjuvant in each side after closing skin.
  Interventions: Drug: Hyaluronidase
- Group C (Placebo Comparator): patients will received TAB block with 19 ml bupivacaine 0.25 % plus 1 ml 0.9% normal saline without any adjuvant in each side after closing skin.
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Hyaluronidase — hyaluronidase will be applied as adjuvant to bupivacaine in transversus abdominis plane block to enhance the postoperative analgesic effect after CS
  Arms: Group H1; Group H2
Drug: Bupivacaine Injection — 20ml bupivacaine will be injected without additives in the transversus abdominis plane block on each side for postoperative analgesic after CS
  Arms: Group C

SUMMARY:
Since TAP block needs to affect several nerves in single tissue plane with a single prick, hyaluronidase is expected to aid greatly in the spread of the LA and help the block. However, there have not been adequate studies to establish the efficacy of adding hyaluronidase in lateral TAP after cesarean section. Hence, the present study was carried out to evaluate the efficacy of hyaluronidase in different concentrations added to bupivacaine in US-guided bilateral lateral TAP block.

ELIGIBILITY:
Inclusion Criteria:

* parturients who aged between 18-40 years old
* with ASA physical status grade II and
* scheduled for elective CS under spinal anesthesia

Exclusion Criteria:

* patients with ASA grade III or IV,
* refusal to participate,
* emergency CS or complicated pregnancy,
* those with bleeding disorders or on anticoagulants,
* those with severe respiratory and cardiovascular diseases,
* having any local infection at the injection site,
* history of allergy to one of the used drugs,
* obese patients (body mass index ≥ 30 kg/m2).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
the duration of analgesia | 24 hours postoperative
  the interval between performing the block and the time of the first request for analgesia.

SECONDARY OUTCOMES:
the postoperative pain severity | every 0,2,4,8,12, up to 24 hours postoperative
  pain was assessed by the visual analog scale (VAS) pain score (range, 0-10; 0, no pain; 10, worst pain)
total morphine consumption | at 24 hours postoperatively
patient satisfaction | at 24 hours postoperatively
  assessed on a four-point scale (1, excellent; 2, good; 3, fair; 4, poor)

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No